CLINICAL TRIAL: NCT07372807
Title: Safety and Efficacy of Ripertamab in Generalized Myasthenia Gravis
Brief Title: Ripertamab for the Treatment of Myasthenia Gravis
Acronym: RIPERT-MG
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Zhongming Qiu (Other)
Responsible Party: Sponsor-Investigator, Zhongming Qiu, Professor, Xinqiao Hospital of Chongqing
Organization: Xinqiao Hospital of Chongqing (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-426
Record Dates: First submitted 2026-01-19; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Myasthenia Gravis (MG)
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental)
  Interventions: Drug: ripertamab

INTERVENTIONS:
Drug: ripertamab — On Day 1 of the treatment period, an intravenous infusion of Ripertamab at a dose of 375 mg/m² body surface area will be administered.
  Other Name:

SUMMARY:
The goal of this clinical trial is to learn if ripertamab works to treat myasthenia gravis. It will also learn about the safety of ripertamab. The main questions it aims to answer are:Will ripertamab improve the symptoms of participants?What medical problems do participants have when using ripertamab?Researchers will compare ripertamab to a placebo (a look-alike substance that contains no drug) to see if ripertamab works to treat chronic inflammatory demyelinating polyneuropathy.Participants will:A single intravenous infusion of ripertamab.Visit the clinic for checkups and tests during W1, W2, W4, W8, W12. Keep a diary of their symptoms and the number of times they undergo rescue therapy.

ELIGIBILITY:
Inclusion Criteria:

(1) Aged ≥ 18 years and ≤ 75 years at screening.(2) Confirmed diagnosis of generalized myasthenia gravis (gMG).(3) Positive for anti-acetylcholine receptor (anti-AChR), anti-muscle-specific kinase (anti-MuSK), and/or anti-low-density lipoprotein receptor-related protein 4 (anti-LRP4) antibodies.(4) A score of ≥ 6 on the Myasthenia Gravis Activities of Daily Living (MG-ADL) Scale, with the ocular subscore accounting for less than 50% of the total score.(5) Classified as Myasthenia Gravis Foundation of America (MGFA) Clinical Classification Types Ⅱ, Ⅲ, or Ⅳ.(6) Voluntary signing of the informed consent form by the patient and/or their legal representative.

Exclusion Criteria:

(1) Any condition that the investigator deems likely to interfere with the evaluation of the study drug, assessment of patient safety, or interpretation of study results.(2) A history of any uncontrolled active infection or severe infection within 8 weeks prior to screening.(3) Receipt of rituximab or any B-cell depleting agent within 6 months prior to screening; note: Subjects with CD19+ or CD20+ B-cell counts above the lower limit of normal are eligible for enrollment.(4) Administration of tocilizumab, eculizumab, mitoxantrone, cyclophosphamide, or other alkylating agents within 3 months prior to the first dose.(5) Administration of immunosuppressants other than glucocorticoids within 1 month prior to the first dose, including but not limited to azathioprine, mycophenolate mofetil, tacrolimus, cyclosporine, and methotrexate.(6) Receipt of plasma exchange (PE), moderate-volume blood transfusion, or immunomodulatory drugs (e.g., interferon β, interferon γ, or intravenous immunoglobulin [IVIG]) within 1 month prior to the first dose.(7) Performance of thymectomy within 12 months prior to baseline, or a planned thymectomy during the 12-week study period.(8) Comorbidity with other chronic active autoimmune diseases requiring treatment with glucocorticoids, biologics, or immunosuppressants (e.g., rheumatoid arthritis, scleroderma).(9) Vaccination with live or attenuated vaccines within 1 month prior to the first dose.(10) A history of previous bone marrow transplantation, hematopoietic stem cell transplantation, total lymphoid irradiation, or T-cell vaccine therapy.(11) Receipt of any investigational drug within 28 days prior to the first dose or 5 times the half-life of the investigational drug, whichever is shorter.(12) Known hypersensitivity to any component of ripertamab.(13) Pregnant or lactating females; for women of childbearing potential (WOCBP) who have not undergone sterilization: refusal to use appropriate contraceptive methods (e.g., oral contraceptives, intrauterine devices [IUDs], or barrier contraception combined with spermicides) from screening until 6 months after the end of treatment.(14) For males who have not undergone sterilization: refusal to use barrier contraception from screening until 6 months after the end of treatment, and refusal to request their partners to use other contraceptive methods (e.g., oral contraceptives, IUDs, barrier methods, or spermicides).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients who achieved a reduction of at least 2 points in the MG-ADL score and did not receive rescue therapy at week 13. | week 13